CLINICAL TRIAL: NCT02897583
Title: A Prospective Randomized Controlled Trial Evaluating the Safety and Efficacy of YAG Vitreolysis Versus Sham for Symptomatic Weiss Ring Due to Posterior Vitreous Detachment
Brief Title: YAG Vitreolysis for Floaters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ophthalmic Consultants of Boston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YAG-001
Record Dates: First submitted 2016-06-16; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Weiss Ring; Floaters; Posterior Vitreous Detachment
MeSH Terms: conditions — vitreous floaters; Vitreous Detachment

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- YAG vitreolysis (Experimental): A Karickoff lens with goniosol will be used to perform the YAG vitreolysis. The number of shots will be determined at the discretion of the treating physician. A focus offset may be used at investigator discretion. Single shot mode will be used. The maximum energy per pulse will be 7 mJ. The endpoint of treatment is the vaporization of the Weiss ring into gas, as well as the disruption of it into smaller fragments as well as any other vitreous opacities deemed visually significant by the treating physician. Only one treatment session will be performed.
  Interventions: Procedure: YAG vitreolysis
- Sham YAG vitreolysis (Sham Comparator): Sham laser treatment will be applied under the same procedure used for laser treatment but by turning the laser power down to 0.3 mJ and using a separate lens covered by a filter that absorbs the power, so no laser enters the eye.
  Interventions: Procedure: YAG vitreolysis

INTERVENTIONS:
Procedure: YAG vitreolysis

SUMMARY:
This is a single-center, prospective randomized controlled trial evaluating the safety and efficacy of YAG vitreolysis versus sham for symptomatic Weiss ring due to posterior vitreous detachment.

DETAILED DESCRIPTION:
52 subjects will be enrolled in the trial and randomized in a 2:1 ratio to receive either YAG laser vitreolysis or sham laser for symptomatic Weiss ring due to posterior vitreous detachment. Subjects will follow up at one week, one month, three months, and six months after the procedure. Assessments will include a questionnaire regarding duration of floater symptoms prior to presentation, severity of floater symptoms, number of floaters, and activity most inconvenienced by presence of floaters; Medical, ocular history and demographics collected; ETDRS and Snellen visual acuity; Optos color photography; Heidelberg Spectralis Optical Coherence Tomography (OCT) and infrared photo; B scan ultrasound of Weiss ring with caliper measurement of nearest distance between Weiss ring and retina, Weiss ring and posterior lens capsule (only in phakic eyes); Slit lamp and indirect ophthalmoscopy with scleral depression of study eye; Applanation tonometry; Visual Functioning Questionnaire-25 (VFQ 25). Qualitative change in Optos photography will evaluated by a masked physician.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of floaters that correlate to the presence of a posterior vitreous detachment for at least 6 months
2. Documented posterior vitreous detachment on clinical examination, OCT, and B scan
3. Self-rating of visual disturbance by the floaters must be at least 4 on a 0-10 scale, with 0 being no symptoms to 10 being debilitating symptoms.
4. Symptomatic Weiss ring (PVD) must be at least 3 mm away from the retina and 5 mm from the posterior lens capsule of the crystalline lens, as measured on B-scan. For pseudophakic patients, there is no minimum required distance from the intraocular lens.
5. Able to position for the YAG laser procedure.
6. Accept the risks of YAG laser including but not limited to retinal detachment, intraocular hemorrhage, retinal damage, cataract formation, optic nerve damage, inflammation, and irreversible loss of vision.
7. Willing and able to comply with clinic visits and study-related procedures
8. If the patient has two symptomatic eyes, only one eye can be randomized and included in the study.
9. Provide signed informed consent

Exclusion Criteria:

1. Snellen best corrected visual acuity worse than 20/50 in the fellow eye
2. History of retinal tear, retinal detachment, or uveitis in the study eye
3. History of diabetic retinopathy, macular edema, retinal vein occlusion, or aphakia in the study eye
4. History of glaucoma or high intraocular pressure defined as having a history of glaucoma surgery or currently taking two or more topical glaucoma medications in the study eye

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2015-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Subjective improvement in floater symptoms | 6 Months
  Questionnaire which asks: "Please rate your visual disturbance by the floaters on a 0-10 scale, with 0 being no symptoms to 10 being debilitating symptoms," "Please quantify your post-operative improvement as a percentage," and "How would you describe your floaters today compared to right before the laser procedure?"

SECONDARY OUTCOMES:
Best Corrected Visual Acuity | 6 Months
  Mean change in visual acuity from Baseline as measured by ETDRS vision testing at 6 months
VFQ-25 Near Activities | 6 Months
  Mean change in baseline in the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) near activities subscale
VFQ-25 Distance Activities | 6 Months
  Mean change in baseline in the National Eye Institute Visual Functioning Questionnaire-25 (NEI VFQ-25) distance activities subscale
Qualitative changes on infrared and color photography | 6 Months
  Qualitative changes on infrared and color photography
Incidence and severity of ocular and systemic adverse events | 6 Months
  Incidence and severity of ocular and systemic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Chirag P Shah, MD, MPH, Principal Investigator — Attending Physician

REFERENCES:
- [Derived] Shah CP, Heier JS. YAG Laser Vitreolysis vs Sham YAG Vitreolysis for Symptomatic Vitreous Floaters: A Randomized Clinical Trial. JAMA Ophthalmol. 2017 Sep 1;135(9):918-923. doi: 10.1001/jamaophthalmol.2017.2388. PMID 28727887